CLINICAL TRIAL: NCT05591404
Title: Investigating the Effects of Social Stress on Brain Imaging
Acronym: SSBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2206000689
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Social Stress
Keywords: Social Stress; fMRI
MeSH Terms: interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Film + TSST (Experimental): Nature Film + Trier Social Stress Test (TSST)
  Interventions: Behavioral: Trier Social Stress Test (TSST)
- Film Only (No-TSST) (No Intervention): Nature Film Only

INTERVENTIONS:
Behavioral: Trier Social Stress Test (TSST) — Participants randomized to the TSST arm will experience the Trier Social Stress Test.
  Arms: Film + TSST

SUMMARY:
The purpose of this study is to examine whether experiencing a social stressor prior to the collection of neuroimaging measures is associated with differences in brain activation in healthy participants.

DETAILED DESCRIPTION:
Using a randomized, parallel-group study design, this scientific investigation will examine the effect that experiencing the Trier Social Stress Test (TSST), the gold-standard for ethically inducing stress in a controlled laboratory setting, may have on neuroimaging measures of anxiety in healthy subjects. The study will enroll 50 healthy subjects who will be randomized to either experience the TSST or watch a nature film prior to undergoing task-based neuroimaging measures of emotional processing and self-referential processing using functional magnetic resonance imaging (fMRI).

This study will be conducted primarily at Massachusetts Institute of Technology with research and clinical support from Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent.
* Sufficiently fluent in English to participate in the trial.
* Between 18-55 years of age (inclusive).
* Right-hand dominant.
* Current medications are stable for past 30 days (no changes to dose or frequency).
* Negative result on pregnancy test (if female).
* Negative result on urine drug screening.
* Liebowitz Social Anxiety Scale (LSAS <30).

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, psychosis, delusional disorders.
* History of eating disorder within past 6 months.
* History of any traumatic brain injury.
* Currently diagnosed with diabetes mellitus.
* Presence of severe medical illness that would prevent completion of study procedures.
* Presence of significant neurological illness or cognitive dysfunction (e.g.; seizures, dementia).
* History of substance use disorder within past 6 months (other than nicotine and caffeine).
* Use of any cannabis-containing products in past 30 days (CBD or THC).
* Use of benzodiazepines in past 2 weeks.
* Use of alpha- or beta-blockers in the past week.
* History of claustrophobia.
* Contraindications for MRI (e.g.; shrapnel).
* Presence of any other medical condition that, in the investigator's opinion, may interfere with the study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Differences in fMRI BOLD Response | 45 minutes after TSST
  Patterns of brain activation measured as blood-oxygenation-level dependent (BOLD) signals will be assessed using 3.0 Tesla (3T) functional magnetic resonance imaging (fMRI). Several exploratory imaging paradigms, including the emotional face-matching task (EFMT) and the self-referential comment task (SRCT), will be used to examine differences between participants who experience the TSST and those who do not.

SECONDARY OUTCOMES:
Change in Acute Subjective Anxiety | -180 minutes, -15 minutes, -5 minutes, +10 minutes, +20 minutes, +30 minutes
  Subjective anxiety will be assessed with a modified Visual Analog Mood Scale (VAMS) which utilizes a vertical 100 millimeter (mm) bipolar visual scale between two opposing moods consisting of the following word pairs: calm-excited, relaxed-tense, and tranquil-troubled. Total subjective anxiety for each timepoint will be the average distance from the top for the three-question battery. VAMS will be assessed 180 minutes before start of TSST, 15 minutes before start of TSST, 5 minutes before start of TSST during the Anticipation phase, after the Stress Procedures (+10 minutes after start of TSST), after 5 minutes in the Recovery Phase (+20 minutes after start of TSST), and 15 minutes after start of the Recovery Phase (+30 minutes after start of TSST).
Differences in Salivary Alpha Amylase | -180 minutes, -15 minutes, -5 minutes, +10 minutes, +20 minutes, +30 minutes
  Physiological stress will be assessed indirectly with salivary alpha amylase (sAA) activity which is regulated by the sympathetic branch of the autonomic nervous system. Samples will be collected using the SalivaBio Oral Swab (SOS) from Salimetrics. Participants will place the SOS in their mouth for 1-2 minutes at each timepoint to collect saliva. sAA will be assessed 180 minutes before start of TSST, 15 minutes before start of TSST, 5 minutes before start of TSST during the anticipation phase, after the Stress Procedures (+10 minutes after start of TSST), after 5 minutes in the Recovery Phase (+20 minutes after start of TSST), and 15 minutes after start of the Recovery Phase (+30 minutes after start of TSST).

CONTACTS AND LOCATIONS:
Overall Officials: John Gabrieli, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data, code, and materials used in the analyses will be made available upon request by John Gabrieli and Massachusetts Institute of Technology after scientific review and a completed data use agreement/material transfer agreement beginning one year after publication of the results. Any requests should be submitted to John Gabrieli at gabrieli@mit.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available beginning one year after publication of the results.
Access Criteria: Data will be provided pending a scientific review and a completed data use agreement/material transfer agreement. Requests should be submitted to John Gabrieli at gabrieli@mit.edu.

REFERENCES:
- See also: SSBI Recruitment Site — https://redcap.link/SSBI